CLINICAL TRIAL: NCT07032272
Title: A Phase 1, Open-label Study to Investigate the Pharmacokinetics and Safety of Remibrutinib (LOU064) in Participants With Severe Renal Impairment Compared to Matched Healthy Participants With Normal Renal Function
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Remibrutinib in Participants With Severe Renal Impairment Compared to Matched Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOU064A2105
Expanded Access: NCT05170724 (Available)
Record Dates: First submitted 2025-06-19; First posted 2025-06-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune and Chronic Inflammatory Diseases
Keywords: Remibrutinib (LOU064); Renal impairment; PK; Safety; Tolerability
MeSH Terms: conditions — Renal Insufficiency | interventions — remibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with severe renal impairment (Experimental): Participants with severe renal impairment will receive remibrutinib
  Interventions: Drug: remibrutinib
- Healthy participants (Experimental): Matched healthy participants will receive remibrutinib
  Interventions: Drug: remibrutinib

INTERVENTIONS:
Drug: remibrutinib — Tablet with oral route of administration

SUMMARY:
The purpose of this study is to support the development of remibrutinib dosing recommendations for patients with impaired renal function.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized study to evaluate the PK after five administrations of remibrutinib in participants with severe RI compared to matched healthy control participants with normal renal function.The purpose of this study is to support the development of remibrutinib dosing recommendations for patients with impaired renal function.

ELIGIBILITY:
Key Inclusion Criteria:

All participants (Group 1 & 2)

* Male and non-childbearing potential female participants 18 to 75 years of age, inclusive, at Screening.
* Must be a non-smoker or a light smoker who smokes no more than 10 cigarettes (or equivalent, including use of nicotine products) per day, at Screening. Smokers must agree to smoke no more than 5 cigarettes (or equivalent) per day from check-in until after Study Completion evaluations.

Participants with severe RI (Group 1)

* Must weigh at least 50 kg to participate in the study and must have a body mass index (BMI) within the range of 18.0 to 35.0 kg/m2, inclusive, at Screening.
* Seated vital signs must be within the following ranges at Screening and Baseline:

  1. body temperature, 35.0 to 37.5°C, inclusive.
  2. systolic blood pressure, 90 to 159 mmHg, inclusive.
  3. diastolic blood pressure, 60 to 99 mmHg, inclusive.
  4. pulse rate, 50 to 99 bpm, inclusive.
* Have impaired renal function as determined by eGFR using the CKD-EPI Creatinine - Cystatin C equation (2021), in the following group at Screening: severe RI; eGFR <30 mL/min, not requiring dialysis.
* Have stable renal function with no clinically significant change in renal status prior to first dosing of study treatment as determined by the Investigator and is not currently or has not been previously on hemodialysis for at least 1 year. Participants with other stable medical disorders such as controlled diabetes, hyperlipidemia, hypothyroidism, arterial hypertension etc., may be eligible as long as they are considered appropriate for enrollment as determined by the Investigator by past medical history, physical examination, ECG, and clinical laboratory tests at Screening.

Healthy control participants (Group 2)

* Each healthy participant must match the age (± 10 years), body weight (± 20%), race, ethnicity and sex of an individual participant in Group 1.
* Must weigh at least 50 kg to participate in the study and must have a BMI within the range of 18.0 to 35.0 kg/m2 inclusive, at Screening.
* Must be in good health as determined by medical history, physical examination, ECG, vital signs and clinical laboratory tests at Screening.
* Has normal renal function with eGFR greater than or equal to 90 mL/min, determined using the CKD-EPI Creatinine - Cystatin C equation (2021) at Screening. Actual creatinine clearance computed over a 24-hour urine collection may be used in place of or in conjunction with the CKD-EPI Creatinine - Cystatin C equation (2021), at the Investigator's discretion.

Key Exclusion Criteria:

All participants (Group 1 & 2)

* Use of other investigational drugs within 5 half-lives or 30 days prior to first dosing of study treatment, whichever is longer, as far as known.
* History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes.
* Use of prescription drugs, OTC medications, or herbal supplements (within the last 2 weeks prior to first dosing, or use of cannabis/marijuana, within the last 4 weeks prior to initial dosing.
* Participants not willing to abstain from food and beverages known to inhibit or induce CYP3A4 from 7 days prior to first dosing and until their respective EoS visit.
* History or presence of malignancy of any organ system (other than treated localized basal cell or squamous cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years of Screening, regardless of whether there is evidence of local recurrence or metastases.
* History or presence of any ongoing, chronic or recurrent infectious disease (including tuberculosis, atypical mycobacterioses, listeriosis, aspergillosis).
* Participants with a history of bone marrow failure or cytopenia will be excluded from the study.
* Is on immunosuppressant therapy or immunomodulators therapy less than or equal to 4 weeks prior to first dosing.
* Any single parameter of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT) or alkaline phosphatase (ALP) exceeding 1.2 x upper limit of normal (ULN) or greater than or equal to 1.5 x ULN total bilirubin (TBL) OR any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or TBL.
* Known or suspected diagnosis of Gilbert's syndrome.

Participants with severe RI (Group 1)

* Clinically significant abnormal findings in physical examination, ECG, or clinical laboratory evaluations, extending over findings related to the known renal disease.
* Participants having had myocardial infarction < 2 years of Screening are not eligible to participate, participants having had myocardial infarction greater than or equal to 2 years of Screening can be eligible to participate.
* Clinically significant illness within 2 weeks prior to first dosing that may jeopardize safety of the study participant and/or alter the study results as judged by the Investigator.
* Participants with end stage renal disease requiring dialysis.

Healthy control participants (Group 2)

* Any clinical laboratory parameters (e.g. hemoglobin, platelets, leukocytes, neutrophils) outside of local laboratory ranges at Screening unless judged not clinically significant by the Investigator.
* Significant illness which has not resolved within 2 weeks prior to first dosing of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-10-12 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Cmax, ss of remibrutinib in blood | Up to 72 hours postdose
  The maximum (peak) observed concentration following multiple-dose administration
AUCtau,ss of remibrutinib in blood | Up to 72 hours postdose
  The area under the curve (AUC) from time zero to the end of the dosing interval (tau) following multiple-dose administration
Ae0-12h,ss of remibrutinib in urine | Up to 12 hours postdose
  Amount of unchanged drug excreted in the urine collection interval from time zero to 12 hours following multiple-dose administration
CLr,ss of remibrutinib in urine | Up to 12 hours postdose
  Renal clearance following multiple-dose administration

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | From Day 1 to end of study (up to 30 days after last administration of study treatment)
  Number of participants with adverse events and serious adverse events
Plasma protein binding of remibrutinib (unbound fraction) | 1 hour postdose
  Fraction unbound based on protein binding data
Cmax,ss,u of remibrutinib in plasma | Up to 72 hours post dose
  The maximum (peak) observed unbound plasma drug concentration following multiple-dose administration
AUCtau,ss,u of remibrutinib in plasma | Up to 72 hours post dose
  The unbound AUC calculated to the end of a dosing interval (tau) following multiple dose administration
AUClast,ss,u of remibrutinib in plasma | Up to 72 hours post dose
  The AUC from time zero to the last measurable unbound concentration sampling time (tlast) following multiple-dose administration
AUClast,ss of remibrutinib in blood | Up to 72 hours postdose
  The AUC from time zero to the last measurable concentration sampling time
Tmax,ss of remibrutinib in blood | Up to 72 hours postdose
  The time to reach maximum (peak) concentration following multiple-dose administration
T1/2 of remibrutinib in blood | Up to 72 hours postdose
  The elimination half-life associated with the terminal slope
CL/F,ss of remibrutinib in blood | Up to 72 hours postdose
  Oral clearance following multiple-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami LLC, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No